CLINICAL TRIAL: NCT05173766
Title: Effects of Ergonomic Considerations on Musculoskeletal Disorders and Posture in Software Developers.
Brief Title: Ergonomic Considerations on Musculoskeletal Disorders and Posture in Software Developers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/Lhr/20/1041/Hafiz Muhammad
Record Dates: First submitted 2021-12-01; First posted 2021-12-30 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ergonomic Principals (Experimental): Ergonomic Principal for computer users will be used.
  Interventions: Other: ergonomic principls

INTERVENTIONS:
Other: ergonomic principls — Ergonomic principles for posture correction in office for computer users.

SUMMARY:
The human and computer interface is becoming increasingly intuitive, but for the inexperienced user still poses formidable problems. Musculoskeletal symptoms of VDU users are believed to have a multifactorial aetiology. Software developers don't have knowledge of ergonomic principles. Faulty postures had an effect on posture.

DETAILED DESCRIPTION:
Data will be collected from software developer companies in Lahore at questionnaire include demographic data and data collection tools. The software developer will be guided about basic ergonomic principles and data will be collected at the start of the study and in 2 stages with a 2-week interval. A quasi-experiment study will be used. The sample size will be323 (margin of error 5%, confidence level 95%, population size 2000, and dist. 50%) by Rao software. A convenient sampling technique will be used. Data will be analyzed using SPSS 21 by comparing mean and correlating variables

ELIGIBILITY:
Inclusion Criteria:

* Software engineers who have experience of more than 2 years, in the same company.
* Software engineers with the age less than 40 years and both gender.

Exclusion Criteria:

* Software engineers who had a past history of spine surgery or diseases in the Spine like disc prolapse, discitis, arthritis etc.
* Orthopedically physically challenged
* Pregnant women.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
The Rapid Entire Body Assessment (REBA) | Change from Baseline Rapid Entire Body Assessment at 3 week
  The Rapid Entire Body Assessment (REBA) was developed to "rapidly" evaluate risk of musculoskeletal disorders (MSD) associated with certain job tasks. Change from Baseline Rapid Entire Body Assessment at 3 week
The Nordic Musculoskeletal Questionnaire (NMQ) | Change from Baseline for musculoskeletal disorders Assessment at 3 week.
  The NMQ can be used as a questionnaire or as a structured interview for musculoskeletal disorders. Change from Baseline for musculoskeletal disorders Assessment at 3 week.
Computer Workstations Tool | Change from Baseline Computer Workstations Assessment at 3 week.
  provided by Occupational Safety and Health Administration. Change from Baseline Computer Workstations Assessment at 3 week.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- I leads Software house, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cassidy, S. and P. Eachus, Developing the computer user self-efficacy (CUSE) scale: Investigating the relationship between computer self-efficacy, gender and experience with computers. Journal of educational computing research, 2002. 26(2): p. 133-153.
- [Background] Punnett L, Wegman DH. Work-related musculoskeletal disorders: the epidemiologic evidence and the debate. J Electromyogr Kinesiol. 2004 Feb;14(1):13-23. doi: 10.1016/j.jelekin.2003.09.015. PMID 14759746
- [Background] Wahlstrom J. Ergonomics, musculoskeletal disorders and computer work. Occup Med (Lond). 2005 May;55(3):168-76. doi: 10.1093/occmed/kqi083. PMID 15857896